CLINICAL TRIAL: NCT00070252
Title: Phase Ib/II Neoadjuvant Trial of the Farnesyltransferase Inhibitor, R115777 With Docetaxel and Capecitabine for Patients With Stage IIIA or IIIB Breast Cancer
Brief Title: Neoadjuvant Tipifarnib, Docetaxel, and Capecitabine in Treating Patients With Locally Advanced or Metastatic Solid Tumors or Stage IIIA or Stage IIIB Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01442; NCI-2012-01442 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WSU-C-2679; MAYO-MC0131; NCI-5599; CDR0000331694; MC0131 (Other: Mayo Clinic); 5599 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2012-12

CONDITIONS: Adult Solid Neoplasm; Inflammatory Breast Carcinoma; Male Breast Carcinoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms, Male; Breast Neoplasms | interventions — Capecitabine; Docetaxel; tipifarnib

ARMS (1):
- Treatment (tipifarnib, capecitabine, docetaxel) (Experimental): Phase Ib: Patients receive oral tipifarnib twice daily and oral capecitabine twice daily on days 1-14 and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Phase II: Patients receive oral tipifarnib twice daily for 6 days. Beginning at least 48 hours after completion of the initial dose of tipifarnib, patients receive treatment as in phase Ib for up to 6 courses at the MTD of capecitabine.
  Interventions: Drug: Capecitabine; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tipifarnib

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Tipifarnib — Given orally (PO)
  Other Names: R115777; Zarnestra

SUMMARY:
Phase I/II trial to study the effectiveness of neoadjuvant tipifarnib combined with docetaxel and capecitabine in treating patients who have locally advanced or metastatic solid tumors or stage IIIA or stage IIIB breast cancer. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy, such as docetaxel and capecitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining tipifarnib with docetaxel and capecitabine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended dose of capecitabine in combination with docetaxel and tipifarnib in patients with locally advanced or metastatic solid tumors. (Phase Ib) II. Determine the complete pathological and clinical response rate in patients with stage IIIA or IIIB breast cancer treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. II. Determine disease-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of capecitabine. Patients in phase II are stratified according to type of breast cancer (inflammatory vs noninflammatory).

Phase Ib: Patients receive oral tipifarnib twice daily and oral capecitabine twice daily on days 1-14 and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive oral tipifarnib twice daily for 6 days. Beginning at least 48 hours after completion of the initial dose of tipifarnib, patients receive treatment as in phase Ib for up to 6 courses at the MTD of capecitabine. Patients in phase Ib are followed at 3 months.

Patients in phase II are followed every 4 months for up to 5 years.

PROJECTED ACCRUAL: A total of 24-53 patients (9-18 for phase Ib and 15-35 for phase II) will be accrued for this study within 14-35 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor

  * Locally advanced or metastatic
* No known standard therapy that is potentially curative or definitely capable of extending life expectancy
* No history of metastatic brain disease within the past 6 months

  * Treated metastatic brain disease is allowed provided disease has been stable for more than 6 months and does not require concurrent steroids or anti-seizure medication
* Histologically confirmed breast cancer

  * Stage IIIA or stage IIIB, including ipsilateral palpable supraclavicular lymph node(s) without other distant metastasis
  * Invasive disease confirmed by 1 of the following*:

    * Incisional biopsy
    * Punch biopsy (applicable for clinical T4b tumors)
    * Core needle (cutting needle) biopsies
* No distant metastatic disease
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-1
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* Bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* AST no greater than 2.5 times ULN
* Creatinine no greater than 1.25 times ULN
* Creatinine clearance at least 50 mL/min
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No diabetes
* No symptomatic neurologic condition
* No other uncontrolled serious medical condition
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of hypersensitivity to intravenous paclitaxel or other medication containing Cremophor EL or polysorbate 80 as a carrier (phase Ib)
* Phase Ib only:

  * More than 4 weeks since prior immunotherapy
  * More than 4 weeks since prior biologic therapy
  * No concurrent immunotherapy
* Phase Ib and II:

  * No concurrent prophylactic filgrastim (G-CSF)
* Phase Ib only:

  * More than 1 year since prior adjuvant docetaxel before metastatic relapse
  * More than 4 weeks since prior chemotherapy and recovered
  * No prior capecitabine AND docetaxel (in combination or as single agents)

    * Prior capecitabine OR docetaxel allowed
  * No other concurrent chemotherapy
* Phase II only:

  * No prior cytotoxic chemotherapy for breast cancer
* Phase Ib only:

  * More than 3 weeks since prior radiotherapy
  * No prior radiotherapy to more than 25% of bone marrow
  * No concurrent radiotherapy
* Phase II only:

  * No prior radiotherapy for breast cancer
* Phase Ib only:

  * More than 4 weeks since prior major surgery
* Phase II only:

  * No prior surgery (other than core or incisional biopsy for diagnostic purposes) for breast cancer
* Phase Ib only:

  * No other ancillary investigational therapy
* Phase Ib and II:

  * No concurrent sorivudine or brivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2003-09; Primary Completion 2006-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (Phase I) | 21 days
Pathologic complete response rate (Phase II) | Up to 5 years
  Estimated by the number of patients with a complete pathologic response divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true pathologic complete response probability will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Clinical tumor response (complete response [CR] or partial response [PR]) (Phase I) | Up to 5 years
  Clinical responses will be summarized by simple descriptive summary statistics.
Overall survival | From registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Toxicity as assessed by the National Cancer Institute (NCI) CTCAE version 3.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Philip, Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Howard University Cancer Center CCOP, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Medical School, Milwaukee, Wisconsin